CLINICAL TRIAL: NCT05825274
Title: Transcranial Direct Current Estimulation for the Treatment of Drug-resistant Epilepsy in Children
Brief Title: TDCs to Treat Drug-resistant Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spanish Foundation for Neurometrics Development (Other)
Responsible Party: Principal Investigator, Moises Domingo, Director Spanish Foundation for Neurometrics Development, Spanish Foundation for Neurometrics Development
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RefEpTDCs
Record Dates: First submitted 2017-09-14; First posted 2023-04-24 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Other Forms of Epilepsy, Treatment Resistant
Keywords: Drug-resistant epilepsy; tDCS
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Intervention Model: Parallel Assignment Masking: Double (Participant, Outcomes Assessor) Primary Purpose: Treatment
Masking Description: we use in half of patient cathodal tDCS or Brain noninvasive stimulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Refractory Epilepsy Group (Experimental): 50 patients with at least they have 3 crisis per week They Receive Cathodal tDCS We do EEG before and after intervention with 19 channels and the patient complete questionnarie: QUALITY OF LIFE IN EPILEPSY - QOLIE-31
  Interventions: Device: Cathodal tDCS
- Placebo Patients (Placebo Comparator): 50 patients with at least they have 3 crisis per week that receive SHAM They Not Receive Cathodal tDCS. We do EEG before and after intervention with 19 channels and the patient complete questionnarie: QUALITY OF LIFE IN EPILEPSY - QOLIE-31
  Interventions: Device: Cathodal tDCS

INTERVENTIONS:
Device: Cathodal tDCS — We do 2 sessions per week of 35 minutes with cathodal electrodes over epileptic focus
  Other Names: Brain Noninvasive Electrical Stimulation; tDCS

SUMMARY:
Epilepsy is the fourth overall neurologic disorder, regardless of age and gender. It encompass a wide spectrum of conditions, intensities and seizure types; therefor, several drugs have proven to treat different types of seizures. However, around 22.5 % of patients are unable to attain control regardless of the drug used or even a combination of several of them. TDCs offers a non-invasive approach with a focal effect for those patients. The focus of this study is to define the role for tDCS in the treatment of drug-resistant epilepsy on children.

DETAILED DESCRIPTION:
Epilepsy is the fourth overall neurologic disorder, regardless of age and gender. There are between 16 and 51 new cases per 100 000 people every year. A community-based study conducted in France concluded that up to 22.5 % of patients could be classified as presenting drug-resistant epilepsy. This group presents significant hazards such as an increased risk of death, injuries, psychosocial disfunction and a reduced quality of life. The International League against Epilepsy defines drug-resistant epilepsy as follows: A failure of adequate trials of two (or more) tolerated, appropriately chosen, appropriately used antiepileptic drugs (whether administered as monotherapies or in a combination) to achieve freedom from seizures. This significant amount of patients are the drive to develop different approaches in order to offer alternatives for control. In this regard, non-invasive brain stimulation protocols lead the way, since the pathophysiological substrate of epilepsy is an enhanced cortical excitability, leading to paroxysmal depolarisation shifts, an enhanced probability of high-frequent and hypersyncronous activity of small neuronal networks and the abnormal spreading of this pathological activity along cortico-cortical and cortico-subcortical neuronal conections. Transcranial direct current stimulation (tDCS) consists of short-lasting electric stimulus delivered to specific brain regions. When delivered repidetly, it generates long-lasting cortical excitability alterations and thus, has the potential to treat epilepsy targeting to the specific brain region where the cortical excitability is alterated. The aim of this study is to define the role for tDCS on the treatment of drug resistant epilepsy on children.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 montths
* Having tried at least two appropriate anti-epileptic drugs (AEDs) tested to tolerance or to blood levels at upper end of the target range of which at least 2 have been tolerated at normal dose.
* At least 2-3 seizure per month documented with EEG, not only clinically.
* In good health except epilepsy.
* Patients or his(her) familys could understand this method and sign the informed consent 7）Patients with good compliance and could complete postoperative follow-up.

Exclusion Criteria:

* Results of MRI remind epilepsy caused by intracranial space-occupying lesions.
* Tumor, cardiopulmonary anomaly, progressive neurological diseases, asthma，mental disease，pepticulcer，diabetes Type 1，bad health etc, and other surgical contraindication
* sleep-related breathing disorders

Ages: 18 Months to 120 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
Decrease in number of crisis per day | 4 months
  Improve epilepsy and EEG (NO statistically and clinically significant spikes or slow waves were observed in EEG)., and changes in scale: QUALITY OF LIFE IN EPILEPSY - QOLIE-31
Body mass index | 4 Months
  kg / m^2

SECONDARY OUTCOMES:
Quality live improve | 4 months
  less drugs consum and number of crisis per week, or moderate changes in EEG or brainwaves
Kessler Foundation Neglect Assessment Process | 4 Months
  During each assessment session, occupational therapists measured patients' functions with the KF-NAP, Functional Independence Measure (FIM™) and Barthel Index (BI)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Neville, MD, Study Director — New Remedies Ltd
Locations (1):
- New Remedies Ltd, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
neuroterapias.es is the database where our foundation recorda all the clinical data of our assays
Supporting Information: ICF, CSR
Time Frame: 4 Months
Access Criteria: login and password previous registration in neuroterapias.es
URL: http://www.neuroterapias.es/

REFERENCES:
- [Result] Varga ET, Terney D, Atkins MD, Nikanorova M, Jeppesen DS, Uldall P, Hjalgrim H, Beniczky S. Transcranial direct current stimulation in refractory continuous spikes and waves during slow sleep: a controlled study. Epilepsy Res. 2011 Nov;97(1-2):142-5. doi: 10.1016/j.eplepsyres.2011.07.016. Epub 2011 Aug 31. PMID 21885255
- [Result] Strzelczyk A, Griebel C, Lux W, Rosenow F, Reese JP. The Burden of Severely Drug-Refractory Epilepsy: A Comparative Longitudinal Evaluation of Mortality, Morbidity, Resource Use, and Cost Using German Health Insurance Data. Front Neurol. 2017 Dec 22;8:712. doi: 10.3389/fneur.2017.00712. eCollection 2017. PMID 29312132
- [Result] Engel J Jr. Approaches to refractory epilepsy. Ann Indian Acad Neurol. 2014 Mar;17(Suppl 1):S12-7. doi: 10.4103/0972-2327.128644. PMID 24791078